CLINICAL TRIAL: NCT01852604
Title: A Randomized Study to Evaluate the Safety and Efficacy of IDX719 in Combinations With Simeprevir and/or TMC647055/Ritonavir With or Without Ribavirin for 12 Weeks in Subjects With Chronic Hepatitis C Infection
Brief Title: Samatasvir (IDX719) in Combinations With Simeprevir and/or TMC647055/Ritonavir With or Without Ribavirin for 12 Weeks in Participants With Chronic Hepatitis C Infection (MK-1894-005)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1894-005; IDX-06A-005 (Other: Idenix Protocol Number)
Record Dates: First submitted 2013-05-06; First posted 2013-05-14 (Estimated); Last update posted 2015-04-23 (Estimated); Status verified 2015-04

CONDITIONS: Chronic Hepatitis C Virus
Keywords: HCV; Hepatitis C; chronic hepatitis C; antiviral
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C | interventions — samatasvir; Simeprevir; Ribavirin; 27-cyclohexyl-12,13,16,17-tetrahydro-22-methoxy-11,17-dimethyl-10,10-dioxide-2,19-methano-3,7:4,1-dimetheno-1H,11H-14,10,2,9,11,17-benzoxathiatetraazacyclo docosine-8,18(9H,15H)-dione; Ritonavir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- Part A: GT 1b, 4 - samatasvir 50/simeprevir/RBV (Experimental): Part A: Participants with genotype 1b or 4 received samatasvir 50 mg and samatasvir matching placebo once daily, plus simeprevir 150 mg capsule once daily, plus RBV (dosing weight-based, according to product label) twice daily for 12 weeks
  Interventions: Drug: Samatasvir; Drug: Simeprevir; Drug: Ribavirin (RBV); Biological: Pegylated interferon (Peg-IFN); Other: Samatasvir matching placebo
- Part A: GT 1b, 4 - samatasvir 100/simeprevir/RBV (Experimental): Part A: Participants with genotype 1b or 4 received samatasvir 100 mg and samatasvir matching placebo once daily, plus simeprevir 150 mg capsule once daily, plus RBV (dosing weight-based, according to product label) twice daily for 12 weeks
  Interventions: Drug: Samatasvir; Drug: Simeprevir; Drug: Ribavirin (RBV); Biological: Pegylated interferon (Peg-IFN); Other: Samatasvir matching placebo
- Part A: GT 1b, 4 - samatasvir 150/simeprevir/RBV (Experimental): Part A: Participants with genotype 1b or 4 received samatasvir 150 mg once daily, plus simeprevir 150 mg capsule once daily, plus RBV (dosing weight-based, according to product label) twice daily for 12 weeks
  Interventions: Drug: Samatasvir; Drug: Simeprevir; Drug: Ribavirin (RBV); Biological: Pegylated interferon (Peg-IFN)
- Part B: GT 1b, 4 - samatasvir 25/simeprevir/RBV (Experimental): Part B: Participants with genotype 1b or 4 received samatasvir 25 mg once daily, plus simeprevir 150 mg capsule once daily, plus RBV (dosing weight-based, according to product label) twice daily for 12 weeks
  Interventions: Drug: Samatasvir; Drug: Simeprevir; Drug: Ribavirin (RBV); Biological: Pegylated interferon (Peg-IFN)
- Part B: GT 1b, 4 - samatasvir 100/simeprevir/RBV (Experimental): Part B: Participants with genotype 1b or 4 received samatasvir 100 mg once daily, plus simeprevir 150 mg capsule once daily, plus RBV (dosing weight-based, according to product label) twice daily for 12 weeks
  Interventions: Drug: Samatasvir; Drug: Simeprevir; Drug: Ribavirin (RBV); Biological: Pegylated interferon (Peg-IFN)
- Part B: GT 6 - samatasvir 100/simeprevir/RBV (Experimental): Part B: Participants with Genotype 6 received samatasvir 100 mg once daily, plus simeprevir 150 mg capsule once daily, plus RBV (dosing weight-based, according to product label) twice daily for 12 weeks
  Interventions: Drug: Samatasvir; Drug: Simeprevir; Drug: Ribavirin (RBV); Biological: Pegylated interferon (Peg-IFN)
- Part C: GT 1a, 1b - samatasvir 50/simeprevir/TCM647055/RTV (Experimental): Part C: Participants with Genotype 1a or 1b received samatasvir 50 mg once daily, plus simeprevir 75 mg capsule once daily, plus TMC647055 450 mg once daily plus RTV 30 mg once daily for 12 weeks
  Interventions: Drug: Samatasvir; Drug: Simeprevir; Drug: Ribavirin (RBV); Drug: TMC647055; Drug: Ritonavir (RTV); Biological: Pegylated interferon (Peg-IFN)
- Part C: GT 1a, 1b - samatasvir 50/simeprivir/TCM647055/RTV/RBV (Experimental): Part C: Participants with Genotype 1a or 1b received samatasvir 50 mg once daily, plus simeprevir 75 mg capsule once daily, plus TMC647055 450 mg once daily, plus RTV 30 mg once daily, plus RBV (dosing weight-based, according to product label) twice daily for 12 weeks
  Interventions: Drug: Samatasvir; Drug: Simeprevir; Drug: Ribavirin (RBV); Drug: TMC647055; Drug: Ritonavir (RTV); Biological: Pegylated interferon (Peg-IFN)

INTERVENTIONS:
Drug: Samatasvir — Samatasvir (IDX719) will be supplied as 25 mg and 50 mg oral tablets.
Drug: Simeprevir — Simeprevir will be supplied as 75 and 150 mg oral capsules.
Drug: Ribavirin (RBV) — Ribavirin will be supplied as 200 mg oral tablets. Participants in the RBV-free arms experiencing non-response or virologic breakthrough during the treatment period will be offered RBV dosed according to the product label as an add-on to the participant's randomized treatment assignment.
Drug: TMC647055 — TMC647055 will be supplied as 150 mg oral capsules.
  Arms: Part C: GT 1a, 1b - samatasvir 50/simeprevir/TCM647055/RTV; Part C: GT 1a, 1b - samatasvir 50/simeprivir/TCM647055/RTV/RBV
Drug: Ritonavir (RTV) — Ritonavir will be supplied as 80 mg/mL oral solution.
  Arms: Part C: GT 1a, 1b - samatasvir 50/simeprevir/TCM647055/RTV; Part C: GT 1a, 1b - samatasvir 50/simeprivir/TCM647055/RTV/RBV
Biological: Pegylated interferon (Peg-IFN) — Participants experiencing non-response or virologic breakthrough during the treatment period will be offered Peg-IFN (subcutaneous injection) dosed according to the product label as an add-on to the participant's randomized treatment assignment.
Other: Samatasvir matching placebo — Samatasvir matching placebo will be supplied for the 50 mg tablets used in Part A.
  Arms: Part A: GT 1b, 4 - samatasvir 100/simeprevir/RBV; Part A: GT 1b, 4 - samatasvir 50/simeprevir/RBV

SUMMARY:
Parts A and B of this study are designed to evaluate the safety, tolerability, efficacy and pharmacokinetic profiles of samatasvir and simeprevir when administered in combination with ribavirin (RBV) for 12 weeks in treatment-naïve, Genotype (GT) 1b, 4 and 6 hepatitic C virus (HCV)-infected participants.

Part C of this study is designed to evaluate the safety, tolerability, efficacy and pharmacokinetic profiles of samatasvir, simeprevir, TMC647055 and ritonavir (RTV) when administered in combination with or without RBV for 12 weeks in treatment-naïve or interferon/RBV-treatment relapsed, GT 1a and 1b HCV-infected participants.

DETAILED DESCRIPTION:
Part A of this study is randomized and double-blind. Parts B and C are randomized and open-label.

ELIGIBILITY:
Inclusion Criteria:

* Must have Genotype 1a, 1b, 4 or 6 HCV infection.
* Documented clinical history compatible with chronic hepatitis C
* HCV treatment-naïve or interferon/RBV-treatment relapsed (Part C)
* Must agree to use an acceptable double method of birth control (one of which must be a barrier method) for at least 6 months after the last dose of study drugs.

Exclusion Criteria:

* Female participants who are pregnant or breastfeeding.
* Body Mass Index (BMI) > 36 kg/m2.
* Co-infected with hepatitis B virus or human immunodeficiency virus (HIV).
* History of hepatocellular carcinoma (HCC) or findings suggestive of possible HCC.
* History or signs of decompensated liver disease: ascites, variceal bleeding, hepatic encephalopathy, spontaneous bacterial peritonitis, or other clinical signs of portal hypertension or hepatic insufficiency.
* Has one or more known primary or secondary causes of liver disease, other than hepatitis C
* History of, or active, acute or chronic, liver or biliary injury due to drugs, toxins, non-HCV viral hepatitis, gallstones or other etiologies
* Donated blood or had significant blood loss 30 days prior to dosing

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2013-03; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Percentage of participants who experienced an adverse event (AE) | Up to approximately 95 weeks
Percentage of participants who experienced a serious adverse event (SAE) | Up to approximately 95 weeks
Percentage of participants who experienced a Grade 1-4 laboratory abnormality | Up to 66 weeks
Percentage of participants who experienced sustained virologic response 4 weeks after the end of treatment (SVR4) | Up to 16 weeks

SECONDARY OUTCOMES:
Percentage of participants who experienced rapid virologic response (RVR) | Week 4
Percentage of participants who experienced early virologic response (EVR) | Week 12
Percentage of participants who experienced sustained virologic response 8 weeks after the end of treatment (SVR8) | Up to 20 weeks
Percentage of participants who experienced sustained virologic response 12 weeks after the end of treatment (SVR12) | Up to 24 weeks
Percentage of participants who experienced sustained virologic response 24 weeks after the end of treatment (SVR24) | Up to 36 weeks
Pharmacokinetic Parameter:Area under the concentration-time curve from time zero to t | Days 1, 4, 7, 10, 14, 21, 28, 42, 56 and 84
Pharmacokinetic Parameter: Maximum observed drug concentration (Cmax) | Days 1, 4, 7, 10, 14, 21, 28, 42, 56 and 84
Pharmacokinetic Parameter: Trough drug concentration (Ctrough) | Days 1, 4, 7, 10, 14, 21, 28, 42, 56 and 84

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC